CLINICAL TRIAL: NCT00883961
Title: Exercise Following Autologous Peripheral Blood Stem Cell Transplantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Dr. Fernando Dimeo, Dept. of Sports Medicine, Charité Universitätsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EA4/029/09
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Hematological Disease
Keywords: High-dose chemotherapy; Hematological neoplasties; Fatigue; Cancer; Exercise; Sport; Hematologic neoplastic disorders
MeSH Terms: conditions — Hematologic Diseases; Fatigue; Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised exercise (Experimental)
  Interventions: Other: Supervised exercise
- Control group (No Intervention): The patients will not carry out a structured exercise program.

INTERVENTIONS:
Other: Supervised exercise — The patients will carry out a daily endurance exercise program consisting of walking on a treadmill for 30 minutes at an intensity of about 80% of the maximum heart rate under supervision from study personnel.
  Arms: Supervised exercise

SUMMARY:
The study evaluates the effects of a supervised exercise program on the physical performance, the mood and the complications of therapy in patients undergoing a high-dose chemotherapy followed by an autologous peripheral blood stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Hematological disease
* Treatment with high-dose chemotherapy followed by autologous stem cell transplantation
* Understanding of written German

Exclusion Criteria:

* Cardiorespiratory, metabolical, osteoarticular or immunological diseases which can be aggravated by exercise
* Pathological stress-ECG at admission

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-04 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
VO2max | At recruitment and after 3 weeks

SECONDARY OUTCOMES:
Mood | At recruitment and after 3 weeks
Duration of aplasia | 3 weeks
Complications during hospitalization | 3 weeks
Need for transfusion of platelets and red blood cells | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Dimeo, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Section Sports Medicine, Charité Universitätsmedizin Berlin, Hindenburgdamm 30, Berlin, State of Berlin, Germany